CLINICAL TRIAL: NCT00795080
Title: Dynamic Magnetic Resonance Imaging (MRI) and Quantitative MR Cerebral Spinal Fluid (CSF) Flow Studies in Craniovertebral Junction Anomalies
Brief Title: Dynamic MRI and Quantitative MR CSF Flow Studies in Craniovertebral Junction Anomalies
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jayapalli Rajiv Bapuraj, MD, Principal Investigator, University of Michigan
Other Study IDs: HUM 18481
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chiari Malformations
Keywords: CVJ malformations
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Normal volunteers who do not have malformations in their cerebral spinal fluid (CSF)
  Interventions: Procedure: Dynamic cervical MRI scans
- 2: Patients with incidentally discovered Chiari 1 DVS malformation of the cerebral spinal fluid (CSF)
  Interventions: Procedure: Dynamic cervical MRI scans
- 3: Patients with known Chiari or any other CVJ malformations undergoing a workup prior to surgery. Research images will be added to the clinically ordered exams ordered at 3 months and 1 year after surgery.
  Interventions: Procedure: Dynamic cervical MRI scans

INTERVENTIONS:
Procedure: Dynamic cervical MRI scans — Serial MRI examination with the neck in flexion and extension to document changes in the cord compression and cerebral spinal fluid (CSF)

SUMMARY:
The purpose of this study is to decide which position of the neck affects cerebral spinal fluid (CSF) flow between the spinal cord and the brain. CSF is a fluid that flows up and down your spinal cord, around the brain and into the ventricles of the brain.

This study will be done with patients who have abnormalities of the neck, including Chiari 1 malformations.

DETAILED DESCRIPTION:
In this study, subjects will have a dynamic cervical magnetic resonance imaging (MRI) of the craniovertebral junction (CVJ) coupled with CSF flow studies. The studies will assess changes in CSF flow velocities that are associated with with changing position of the neck at the CVJ and aqueduct of Sylvius.

Eligible patients include those with Chiari 1 malformations and similar malformations to the CVJ. This malformation lead to inherent instability in this region and symptoms such as headaches, dizziness, neck pain and other neurological problems. This study will determine if there is any correlation of these MRI findings to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers must be 18 yrs of age or older.
* Patients w/Chiari 1 or CVJ malformations aged 12 yrs or older,
* Able to cooperate in flexing and extending their neck within the cervical spine coil used for MR Imaging.
* Pediatric patients will be included only if they can cooperate for additional sequences done for the study who don't require sedation or any form of anesthesia.

Exclusion Criteria:

* Patients who are medically unstable or cannot voluntarily flex or extend their necks.
* Patients who have hardware in the head or necks which are incompatible with MR imaging.
* Patient requiring any form of sedation which can lead to compromise of the airway with maneuvers described above.
* History of prior head trauma or history of neurological conditions which can result in altered CSF dynamics.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pilot group consisting of 10 healthy volunteers. Patients recruited w/incidental findings of Chiari 1 malformations and Patients recruited with known Chiari and other CVJ malformations (prior to surgery)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-07-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To compare changes in flow velocities at the CVJ (cranial vertebral junction) and aqueduct of Sylvius w/dynamic imaging in normal controls and in patients with symptomatic and asymptomatic Chiari 1 malformations and similar anomalies. | 1 year

SECONDARY OUTCOMES:
Results from the primary outcome will be correlated with post operative changes in a subset of patients as a predictor for surgical outcomes. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Bapuraj, M.D., MD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No